CLINICAL TRIAL: NCT06104904
Title: Enhancing the Capacity of Pediatric Primary Care Providers: a Pilot Trial of Anxiety Action Plan
Brief Title: Managing Anxiety in Pediatric Primary Care (MAPP)
Acronym: MAPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Golda S. Ginsburg, Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-111SO-2; R34MH129410-01 (NIH)
Record Dates: First submitted 2023-10-18; First posted 2023-10-27 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Anxiety; Anxiety Disorders
Keywords: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Managing Anxiety in Pediatric Primary Care (MAPP) (Experimental): Participants receive approximately 4 sessions of a primary care provider-delivered intervention for reducing youth anxiety symptoms based on exposure therapy.
  Interventions: Behavioral: MAPP
- Enhanced Usual Care (EUC) (Placebo Comparator): Participants receive a list of resources on how to reduce anxiety (e.g., videos, books, etc.).
  Interventions: Behavioral: MAPP

INTERVENTIONS:
Behavioral: MAPP — Behavioral intervention based on exposure therapy strategies.

SUMMARY:
The goal of this clinical trial is to conduct a randomized controlled trial to enhance the capacity of pediatric primary care providers to assist their patients who struggle with anxiety.

The study aims to refine and assess the feasibility of the Anxiety Action Plan (AxAP), a brief intervention to reduce pediatric anxiety, delivered by primary care providers (PCPs) in community pediatric primary care clinics. The goal of the AxAP is to enhance the capacity of PCPs to identify and intervene with anxious youth, which will enhance access to care in general and especially in locations with few mental health specialists. PCPs participating in this study will attend a training, administer the intervention to enrolled youth assigned to the MAPP condition, participate in coaching sessions, and fill out study questionnaires. Families participating in this study will complete evaluations with the study team, receive the intervention from their PCP (if assigned to the MAPP condition), and fill out study questionnaires. Researchers will compare the MAPP intervention to Enhanced Usual Care (EUC; consisting of videos, handouts, and other resources for anxiety reduction) to see the differences, if any, in child outcomes.

DETAILED DESCRIPTION:
Anxiety disorders in youth are: 1) the most prevalent psychiatric illnesses, 2) associated with severe disability, and 3) considered gateway disorders--as they predict a broad range of adult psychiatric and functional problems. Despite the high prevalence and impairment, less than half of anxious youth receive mental health services and access to evidenced-based interventions lags far behind that of less common psychiatric illnesses, such as attention deficit hyperactivity disorder. This application addresses this mental health service gap and responds to NIH's priorities in PAR-MH-21-131: Pilot Effectiveness Trials for Treatment, Preventive and Services Interventions (R34) aimed at testing interventions with previous efficacy in community settings using novel service delivery methods. Specifically, the investigators propose to refine and assess the feasibility of the Anxiety Action Plan (AxAP), a brief intervention to reduce pediatric anxiety, delivered by primary care providers (PCPs; defined here as nurse practitioners, physician assistants, and/or pediatricians) in community pediatric primary care clinics. Primary care settings are ideal for addressing pediatric anxiety specifically because: 1) prevalence rates of excessive anxiety are high in primary care (approximately 10-20%), 2) over 90% of anxious youth report physical complaints (e.g., stomach aches) and are "frequent flyers" in primary care settings, 3) children with, compared to without, medical conditions treated by PCPs are more likely to have elevated anxiety, and 4) PCPs are often the first and only health professional children visit. This study builds on the PI's development and feasibility pilot work with PCPs conducted as part of the NIMH-funded Center for Mental Health in Pediatric Primary Care and with school nurses as part of a Department of Education grant. The AxAP, modeled after the Asthma Action Plan familiar to PCPs, is based on the core element of cognitive behavioral therapy for anxiety (i.e., behavioral exposure), was designed to fit within the short primary care visit (20-30 minutes), can be delivered virtually, is brief (1-4 sessions), and can be billed for as an office visit. Uniquely, and in stark contrast to co-location or integrated models, the goal of the AxAP is to enhance the capacity of PCPs to identify and intervene with anxious youth, which will enhance access to care in general and especially in locations with few mental health specialists. If results of this study are positive, findings would support a large effectiveness trial using an intervention that is ready for dissemination and that could significantly improve clinical care for anxious youth, enhance the capacity of PCPs to identify and reduce anxiety, and lower personal and economic costs associated with pediatric anxiety.

ELIGIBILITY:
Inclusion Criteria for youth:

* 6-17 years of age
* Have elevated anxiety symptoms as indicated by a total Screen for Child Anxiety Rated Disorders score between 20 and 55 based on parent and/or child report

Exclusion Criteria for youth:

* Have a medical or psychiatric condition contraindicating participation (e.g., suicidality) based on clinical interview
* Are receiving psychosocial mental health treatment for anxiety

Inclusion Criteria for PCPs:

* PCPs must have a PA, RN, NP, APRN or MD degree and be at least a part time employee in a primary care setting. There are no other inclusion/exclusion criteria.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression Improvement scale | Youth will be assessed at 2 months (post intervention) and 6 months after eligibility is established.
  Improvement in anxiety symptoms and related functioning since baseline (a score of 1 or 2 is defined as a responder; scores of 3-7 are defined as non-responders).
Primary Care Provider Primary outcome | Post intervention (i.e., 2 months after first family enrolled)
  Satisfaction with MAPP: 70% of PCPs endorsing a score of 3 (somewhat helpful) or higher on a question asking "how helpful they perceived the program to be"; scores range from 0 (not at all helpful) to 4 very helpful.

CONTACTS AND LOCATIONS:
Overall Officials: Golda S Ginsburg, PhD, Principal Investigator — UConn Health
Locations (1):
- UConn Health, West Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
As per NIMH requirements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of primary and secondary outcome results.
Access Criteria: Researchers can request data from PI